CLINICAL TRIAL: NCT05663151
Title: Mechanisms Underlying the Efficacy of Prolonged Exposure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Collaborators: National Center for PTSD (U.S. Federal Agency)
Responsible Party: Principal Investigator, Suzanne Pineles, Principal Investigator/Study Chair, VA Boston Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1577670
Record Dates: First submitted 2022-11-22; First posted 2022-12-23 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Prolonged Exposure Therapy; PTSD; Sleep
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prolonged Exposure Therapy for Posttraumatic Stress Disorder (Experimental): 15 participants who meet study inclusion/exclusion criteria will be individually administered a full course of PE during 10, 60 minute-sessions, with independent multimodal assessment batteries administered at pre-treatment, mid-treatment (post session 5), post-treatment, and a 1-month follow-up.
  Interventions: Behavioral: Prolonged Exposure Therapy for Posttraumatic Stress Disorder

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy for Posttraumatic Stress Disorder — Participation will occur throughout 17 weeks over 15 separate visits during which 10, 60-minute sessions of PE will take place. Session 1 of PE will focus on psychoeducation. Session 2 of PE will involve a continuation of psychoeducation and rationale for exposure as well as the collaborative construction of the in vivo exposure hierarchy. After session 2, participants will begin homework where they are instructed to confront situations on their hierarchy. Starting in session 3 of PE, participants will begin imaginal exposures to their worst trauma memory. This involves the participant recounting and visualizing the trauma memory aloud with the clinician in the room for 30-40 minutes. The session will end with 15-20 minutes of processing the imaginal exposure. Participants will continue in-session imaginal exposures until the end of treatment. Throughout the treatment, participants will listen to a recording of their imaginal exposure and engage in in vivo exposures daily.

SUMMARY:
The primary objective of this research is to collect pilot data that demonstrates that proposed neural, psychophysiological and subjective markers measured before, during, and after treatment change over the course of Prolonged Exposure therapy (PE) for posttraumatic stress disorder (PTSD). The aims of the study are to: (1) examine theoretically informed mechanisms as pre-treatment predictors of PE treatment efficacy, (2) characterize how neural, psychophysiological, and subjective markers measured before, during, and after treatment change over the course of PE, and (3) examine proposed mechanisms of change as measures of PE treatment efficacy. This is a longitudinal study of predictors of exposure therapy efficacy that will be conducted within the context of a standard 10 session PE treatment trial, with independent multimodal assessment batteries administered at pre-treatment, mid-treatment, post-treatment, and at 1-month follow-up. This data will be used to support a future NIMH and/or VA grant submission.

DETAILED DESCRIPTION:
Proposed research sets to collect pilot data to examine how the proposed neural, psychophysiological and subjective markers measured before, during, and after treatment change over the course of Prolonged Exposure (PE) therapy for posttraumatic stress disorder (PTSD). Fifty participants will be screened with the goal of obtaining 15 participants to complete the study. Participants will complete ten 60-minute sessions of PE. During each PE session, participants will be outfitted with a NINscan device to record psychophysiological measures including skin conductance, heart rate, and facial EMG, as well as neural measures of LPFC activity. Multimodal assessment batteries will be scheduled to take place at pre-treatment, mid-treatment (i.e., post session 5), post-treatment (i.e., post-session 10), and at 1-month follow-up. These sessions will include a battery of self-report measures, clinician-administered diagnostic interviews, and script-driven imagery (SDI) procedures with physiologic and neural recordings. The primary outcome measure will be PTSD symptom change on the CAPS-5 and the secondary outcome measures will be a) change in self-reported symptom severity, b) premature treatment dropout, and c) change in psychophysiological reactivity and LPFC activity during the SDI procedures. This proposed research will inform theoretical models of exposure therapy efficacy, with the goal of enhancing prolonged exposure therapy.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of PTSD as defined by DSM-5 (as indicated by meeting diagnostic criteria on the CAPS-5)
2. interest in starting PE (as indicated during the informed consent process)
3. Veteran

Exclusion Criteria:

1. Current or past history of schizophrenic or other psychotic disorders,
2. Untreated Bipolar Disorder or a history of a manic/mixed episode within the last 6 months,
3. Severe traumatic brain injury,
4. Major neurological problems,
5. Current substance use disorder,
6. Active risk to self or others,
7. Current participation in cognitive-behavioral therapy,
8. Previously received > 2 sessions of Prolonged Exposure, and
9. Having no memory of their traumatic event.
10. For participants who are currently prescribed psychotropic medication, they will be eligible for the study provided medication use has been stable for 2 months prior to enrollment and remains stable throughout participation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Clinician Administered PTSD Scale for DSM-5 (CAPS-5) | Given during screening session, pre-treatment, mid-treatment (post session 5 in week 5 of treatment), post-treatment (post session 10 in week 10 of treatment), and at 1-month follow up.
  The primary clinical outcome, CAPS-5, is the gold standard clinical interview for assessing PTSD severity. In CAPS-5, each of the 20 symptoms of PTSD is rated on a 5-point severity scale ranging from 0 (absent) to 4 (extreme). Total scores range from 0 to 80.

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Given during screening session, pre-treatment, mid-treatment (post session 5 in week 5 of treatment), post-treatment (post session 10 in week 10 of treatment), and at 1-month follow up.
  Self-ratings of how much one is bothered by each of the 20 symptoms of PTSD on a 5-point severity scale ranging from 0 (Not at all) to 4 (extremely)
QIDS-SR (93) | Given during screening session, pre-treatment, mid-treatment (post session 5 in week 5 of treatment), post-treatment (post session 10 in week 10 of treatment), and at 1-month follow up.
  Used to measure severity of depressive symptoms. provides equivalent weightings (0-3) for each symptom item, gives clearly stated anchors that estimate the frequency and severity of symptoms, and includes all items required to diagnose a major depressive episode (approximately 5 minutes)
Prefrontal cortical activity during script-driven imagery (SDI) | Given during screening session, pre-treatment, mid-treatment (post session 5 in week 5 of treatment), post-treatment (post session 10 in week 10 of treatment), and at 1-month follow up.
  Prefrontal cortical (PFC) activity will be monitored during SDI procedures using NINscan portable brain and physiologic monitoring system via near infrared spectroscopy (NIRS) of the medial and lateral PFC. NIRS yields concentrations of oxygenated (oxyHb) and deoxygenated (deoxyHb) hemoglobin that can be used to assess cortical activation. Various portions of PFC (e.g. Brodmann areas 10, 46, 44, 45 and 47) have been shown to activate and/or deactivate during script-driven imagery (SDI) of an index trauma in persons with PTSD and to be associated with better PE outcome. NIRS data will be converted to quantitative oxy-Hb, deoxy-Hb, and total-Hb using the modified Beer-Lambert law. Changes in quantitative hemodynamic measure (oxy-Hb, deoxy-Hb, total-Hb) will be compared between 30 s of trauma-related SDI and their baseline epochs (30 s of silence preceding the respective script).
Change in electrocardiography (ECG) and heart rate variability (HRV) during script driven imagery (SDI) | Given during screening session, pre-treatment, mid-treatment (post session 5 in week 5 of treatment), post-treatment (post session 10 in week 10 of treatment), and at 1-month follow up.
  ECG will be monitored during SDI procedures using NINscan portable brain and physiologic monitoring system. ECG will be collected continuously and the relative change calculated by subtracting the average ECG level for the 5 seconds immediately preceding SDI onset from the maximum level within 1 to 5 seconds after SDI onset. Heart rate variability (HRV) will be calculated form 5-minute epochs during baseline, calculating the standard deviation of all NN intervals, and comparing them to 5-minute intervals after onset of SDI. The ECG and HRV signals will be assessed individually and also in combination using posterior probability scores. Changes in ECG and HRV have been shown to indicate differential sympathetic reactivity in persons with PTSD versus controls.
Change in skin conductance (SC) during script-driven imagery (SDI) | Given during screening session, pre-treatment, mid-treatment (post session 5 in week 5 of treatment), post-treatment (post session 10 in week 10 of treatment), and at 1-month follow up.
  SC will be monitored during SDI procedures using NINscan portable brain and physiologic monitoring system. SC level for the 5 seconds immediately preceding SDI onset from the maximum level within 1 to 5 seconds after SDI onset. This response window is selected to reduce the likelihood that response scores would be contaminated by spontaneous SC fluctuations. The signals will be assessed individually and also in combination using posterior probability scores. Changes in SC signals have been shown to indicate differential sympathetic reactivity in persons with PTSD versus controls.
Change in electromyography (EMG) during script-driven imagery (SDI) | Given during screening session, pre-treatment, mid-treatment (post session 5 in week 5 of treatment), post-treatment (post session 10 in week 10 of treatment), and at 1-month follow up.
  Electromyography of the corrugator muscle will be monitored during SDI procedures using NINscan portable brain and physiologic monitoring system. An EMG response (EMGR) score will be calculated by subtracting the average EMG level for the 5 seconds immediately preceding SDI onset from the maximum level during SDI. The signals will be assessed individually and also in combination using posterior probability scores. Changes in corrugator EMG have been shown to indicate differential sympathetic reactivity in persons with PTSD versus controls.
Change in respirometry during script-driven imagery (SDI) | Given during screening session, pre-treatment, mid-treatment (post session 5 in week 5 of treatment), post-treatment (post session 10 in week 10 of treatment), and at 1-month follow up.
  Changes in respirometry will be monitored during SDI procedures using NINscan portable brain and physiologic monitoring system. Average frequency and signal amplitude during baseline and SDI exposure epochs will be compared to calculate the relative change in respirometry. Changes in respirometry have been shown to indicate differential sympathetic reactivity in persons with PTSD versus controls.
Premature treatment dropout | Given at pre-treatment and mid-treatment (post session 5 in week 5 of treatment).
  Maintenance of active participation or dropout from the treatment will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Pineles, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared after study completion.
Supporting Information: Study Protocol
Time Frame: Data will be available within a year of submission after publications.

REFERENCES:
- [Background] Powers MB, Halpern JM, Ferenschak MP, Gillihan SJ, Foa EB. A meta-analytic review of prolonged exposure for posttraumatic stress disorder. Clin Psychol Rev. 2010 Aug;30(6):635-41. doi: 10.1016/j.cpr.2010.04.007. Epub 2010 May 2. PMID 20546985
- [Background] Hembree EA, Foa EB, Dorfan NM, Street GP, Kowalski J, Tu X. Do patients drop out prematurely from exposure therapy for PTSD? J Trauma Stress. 2003 Dec;16(6):555-62. doi: 10.1023/B:JOTS.0000004078.93012.7d. PMID 14690352
- [Background] Schnurr PP, Friedman MJ, Engel CC, Foa EB, Shea MT, Chow BK, Resick PA, Thurston V, Orsillo SM, Haug R, Turner C, Bernardy N. Cognitive behavioral therapy for posttraumatic stress disorder in women: a randomized controlled trial. JAMA. 2007 Feb 28;297(8):820-30. doi: 10.1001/jama.297.8.820. PMID 17327524
- [Background] Kehle-Forbes SM, Meis LA, Spoont MR, Polusny MA. Treatment initiation and dropout from prolonged exposure and cognitive processing therapy in a VA outpatient clinic. Psychol Trauma. 2016 Jan;8(1):107-114. doi: 10.1037/tra0000065. Epub 2015 Jun 29. PMID 26121175
- [Background] Schottenbauer MA, Glass CR, Arnkoff DB, Tendick V, Gray SH. Nonresponse and dropout rates in outcome studies on PTSD: review and methodological considerations. Psychiatry. 2008 Summer;71(2):134-68. doi: 10.1521/psyc.2008.71.2.134. PMID 18573035
- [Background] Bouton ME, Mineka S, Barlow DH. A modern learning theory perspective on the etiology of panic disorder. Psychol Rev. 2001 Jan;108(1):4-32. doi: 10.1037/0033-295x.108.1.4. PMID 11212632
- [Background] McGuire JF, Lewin AB, Storch EA. Enhancing exposure therapy for anxiety disorders, obsessive-compulsive disorder and post-traumatic stress disorder. Expert Rev Neurother. 2014 Aug;14(8):893-910. doi: 10.1586/14737175.2014.934677. Epub 2014 Jun 27. PMID 24972729
- [Background] Rachman S. Emotional processing. Behav Res Ther. 1980;18(1):51-60. doi: 10.1016/0005-7967(80)90069-8. No abstract available. PMID 7369988
- [Background] Wisco BE, Baker AS, Sloan DM. Mechanisms of Change in Written Exposure Treatment of Posttraumatic Stress Disorder. Behav Ther. 2016 Jan;47(1):66-74. doi: 10.1016/j.beth.2015.09.005. Epub 2015 Oct 8. PMID 26763498
- [Background] Pitman RK, Orr SP, Altman B, Longpre RE, Poire RE, Macklin ML, Michaels MJ, Steketee GS. Emotional processing and outcome of imaginal flooding therapy in Vietnam veterans with chronic posttraumatic stress disorder. Compr Psychiatry. 1996 Nov-Dec;37(6):409-18. doi: 10.1016/s0010-440x(96)90024-3. PMID 8932965
- [Background] Robison-Andrew EJ, Duval ER, Nelson CB, Echiverri-Cohen A, Giardino N, Defever A, Norrholm SD, Jovanovic T, Rothbaum BO, Liberzon I, Rauch SA. Changes in trauma-potentiated startle with treatment of posttraumatic stress disorder in combat Veterans. J Anxiety Disord. 2014 May;28(4):358-62. doi: 10.1016/j.janxdis.2014.04.002. Epub 2014 Apr 15. PMID 24786361
- [Background] Craske MG, Kircanski K, Zelikowsky M, Mystkowski J, Chowdhury N, Baker A. Optimizing inhibitory learning during exposure therapy. Behav Res Ther. 2008 Jan;46(1):5-27. doi: 10.1016/j.brat.2007.10.003. Epub 2007 Oct 7. PMID 18005936
- [Background] Hayes, S.C., K.D. Strosahl, and K.G. Wilson, Acceptance and commitment therapy. 2009: American Psychological Association
- [Background] Bryant RA, Felmingham K, Kemp A, Das P, Hughes G, Peduto A, Williams L. Amygdala and ventral anterior cingulate activation predicts treatment response to cognitive behaviour therapy for post-traumatic stress disorder. Psychol Med. 2008 Apr;38(4):555-61. doi: 10.1017/S0033291707002231. Epub 2007 Nov 16. PMID 18005496
- [Background] van Rooij SJ, Geuze E, Kennis M, Rademaker AR, Vink M. Neural correlates of inhibition and contextual cue processing related to treatment response in PTSD. Neuropsychopharmacology. 2015 Feb;40(3):667-75. doi: 10.1038/npp.2014.220. Epub 2014 Aug 26. PMID 25154707
- [Background] Fonzo GA, Goodkind MS, Oathes DJ, Zaiko YV, Harvey M, Peng KK, Weiss ME, Thompson AL, Zack SE, Lindley SE, Arnow BA, Jo B, Gross JJ, Rothbaum BO, Etkin A. PTSD Psychotherapy Outcome Predicted by Brain Activation During Emotional Reactivity and Regulation. Am J Psychiatry. 2017 Dec 1;174(12):1163-1174. doi: 10.1176/appi.ajp.2017.16091072. Epub 2017 Jul 18. PMID 28715908
- [Background] Fonzo GA, Goodkind MS, Oathes DJ, Zaiko YV, Harvey M, Peng KK, Weiss ME, Thompson AL, Zack SE, Mills-Finnerty CE, Rosenberg BM, Edelstein R, Wright RN, Kole CA, Lindley SE, Arnow BA, Jo B, Gross JJ, Rothbaum BO, Etkin A. Selective Effects of Psychotherapy on Frontopolar Cortical Function in PTSD. Am J Psychiatry. 2017 Dec 1;174(12):1175-1184. doi: 10.1176/appi.ajp.2017.16091073. Epub 2017 Jul 18. PMID 28715907
- [Background] McLaughlin AA, Keller SM, Feeny NC, Youngstrom EA, Zoellner LA. Patterns of therapeutic alliance: rupture-repair episodes in prolonged exposure for posttraumatic stress disorder. J Consult Clin Psychol. 2014 Feb;82(1):112-21. doi: 10.1037/a0034696. Epub 2013 Nov 4. PMID 24188510
- [Background] Pace-Schott EF, Germain A, Milad MR. Effects of sleep on memory for conditioned fear and fear extinction. Psychol Bull. 2015 Jul;141(4):835-57. doi: 10.1037/bul0000014. Epub 2015 Apr 20. PMID 25894546
- [Background] Pace-Schott EF, Germain A, Milad MR. Sleep and REM sleep disturbance in the pathophysiology of PTSD: the role of extinction memory. Biol Mood Anxiety Disord. 2015 May 29;5:3. doi: 10.1186/s13587-015-0018-9. eCollection 2015. PMID 26034578
- [Background] Pace-Schott EF, Bottary RM, Kim SY, Rosencrans PL, Vijayakumar S, Orr SP, Lasko NB, Goetter EM, Baker AW, Bianchi MT, Gannon K, Hoeppner SS, Hofmann SG, Simon NM. Effects of post-exposure naps on exposure therapy for social anxiety. Psychiatry Res. 2018 Dec;270:523-530. doi: 10.1016/j.psychres.2018.10.015. Epub 2018 Oct 9. PMID 30340182
- [Background] Lanius RA, Bluhm R, Lanius U, Pain C. A review of neuroimaging studies in PTSD: heterogeneity of response to symptom provocation. J Psychiatr Res. 2006 Dec;40(8):709-29. doi: 10.1016/j.jpsychires.2005.07.007. Epub 2005 Oct 7. PMID 16214172
- [Background] van Rooij SJ, Rademaker AR, Kennis M, Vink M, Kahn RS, Geuze E. Impaired right inferior frontal gyrus response to contextual cues in male veterans with PTSD during response inhibition. J Psychiatry Neurosci. 2014 Sep;39(5):330-8. doi: 10.1503/jpn.130223. PMID 24886789
- [Background] Pineles SL, Suvak MK, Liverant GI, Gregor K, Wisco BE, Pitman RK, Orr SP. Psychophysiologic reactivity, subjective distress, and their associations with PTSD diagnosis. J Abnorm Psychol. 2013 Aug;122(3):635-44. doi: 10.1037/a0033942. PMID 24016006
- [Background] Clark LA, Watson D, Mineka S. Temperament, personality, and the mood and anxiety disorders. J Abnorm Psychol. 1994 Feb;103(1):103-16. PMID 8040472
- [Background] Weathers, F.W., et al., The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). 2012, Interview available from the National Center for PTSD at www.ptsd.va.gov
- [Background] First, M.B., et al., Structured Clinical Interview for DSM-5 Disorders (SCID-5-RV). 2015, Arlington, VA: American Psychiatric Publishing
- [Background] Posner, K., et al., Columbia-suicide severity rating scale (C-SSRS). Columbia University Medical Center, 2008
- [Background] Foa, E., E. Hembree, and B.O. Rothbaum, Prolonged exposure therapy for PTSD: Emotional processing of traumatic experiences therapist guide. 2007: Oxford University Press.
- [Background] Orr SP, Pitman RK, Lasko NB, Herz LR. Psychophysiological assessment of posttraumatic stress disorder imagery in World War II and Korean combat veterans. J Abnorm Psychol. 1993 Feb;102(1):152-9. doi: 10.1037//0021-843x.102.1.152. PMID 8436691
- [Background] Keane TM, Kolb LC, Kaloupek DG, Orr SP, Blanchard EB, Thomas RG, Hsieh FY, Lavori PW. Utility of psychophysiological measurement in the diagnosis of posttraumatic stress disorder: results from a Department of Veterans Affairs Cooperative Study. J Consult Clin Psychol. 1998 Dec;66(6):914-23. doi: 10.1037//0022-006x.66.6.914. PMID 9874904
- [Background] Wechsler, D., WASI-II: Wechsler abbreviated scale of intelligence. 2011: PsychCorp
- [Background] Stern, R.A., et al., The Boston qualitative scoring system for the Rey-Osterrieth complex figure: Description and interrater reliability. The Clinical Neuropsychologist, 1994. 8(3): p. 309-322.
- [Background] Sadeh A. The role and validity of actigraphy in sleep medicine: an update. Sleep Med Rev. 2011 Aug;15(4):259-67. doi: 10.1016/j.smrv.2010.10.001. Epub 2011 Jan 14. PMID 21237680
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Weathers, F.W., et al., The PTSD Checklist for DSM-5 (PCL-5). 2010, Scale available from the National Center for PTSD at www.ptsd.va.gov
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Background] Weathers, F.W., et al., The Life Events Checklist for DSM-5 (LEC-5). 2013: Instrument available from the National Center for PTSD at www.ptsd.va.gov
- [Background] Hatcher, R.L. and J.A. Gillaspy, Development and validation of a revised short version of the working alliance inventory. Psychotherapy Research, 2006. 16(1).